CLINICAL TRIAL: NCT00358397
Title: Phase I Safety Study of Clostridium Novyi-NT Spores in Patients With Treatment-Refractory Solid Tumor Malignancies
Brief Title: One Time Injection of Bacteria to Treat Solid Tumors That Have Not Responded to Standard Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Design Problem
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0590
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Tumors
Keywords: Solid Tumor; Clostridial; Spore-forming bacteria; hypoxia; anaerobes; Clostridium novyi; Bacteria; Bacteriolytic; Tumor lysis; Necrosis; Colon Cancer; Lung Cancer; Sarcoma; Bladder Cancer; Rectal Cancer; Gastric Cancer; Pancreatic Cancer; Experimental Therapy; Solid Tumors
MeSH Terms: conditions — Neoplasms; Hypoxia; Necrosis; Colonic Neoplasms; Lung Neoplasms; Sarcoma; Urinary Bladder Neoplasms; Rectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: Clostridium novyi-NT spores

INTERVENTIONS:
Drug: Clostridium novyi-NT spores

SUMMARY:
This study will include a one time intravenous (IV) infusion of Clostridium novyi-NT (C. novyi-NT) spores to treat solid tumors which have not responded to standard therapy.

DETAILED DESCRIPTION:
Investigators at the SKCCC have developed a bacterial strain (C. novyi-NT) that can infect tumors and destroy them, but does not grow in normal tissues. In animal experiments, a single intravenous injection of these bacteria can cause dramatic regression of many tumors, and the tumors do not recur in approximately (~) 30% of the animals.

This is a phase I dose escalation study using a single dose of Clostridium novyi-NT spores in patients with treatment-refractory solid tumor malignancies. The overall objective of this study is to determine the safety and document any preliminary evidence of anti-tumor activity in this patient population.

ELIGIBILITY:
Inclusion Criteria -

1. Histologically or cytologically proven solid tumor malignancy as proven by referral CT scan of the chest, abdomen and pelvis.
2. Patients must be refractory to standard chemotherapy or for whom no standard treatment exists. At least four weeks must have elapsed since completion of any prior chemotherapy.
3. Patients must have measurable disease; defined as at least one lesion whose longest diameter can be accurately measured as >2 cm.
4. ECOG performance status of 0 or 1.
5. Prior locoregional therapy, including cryotherapy, radiofrequency ablation, or regional chemotherapy is allowed if at least 6 weeks have elapsed.
6. Prior radiation therapy is allowed. At least 6 weeks must have elapsed since the completion of radiation therapy and the patient must have recovered from side effects.
7. Prior systemic radionuclide therapy is allowed. At least 4 weeks must have elapsed since completion of the therapy.
8. Prior surgery is allowed. At least 6 weeks must have elapsed since the completion of major surgery and the patient must be fully recovered from this surgery and any attendant postsurgical complications.
9. Patients must be 18 years of age or older
10. Patients of childbearing potential must use adequate birth control measures (e.g., abstinence, barrier method with spermicide; or use by partner of oral contraceptives, intrauterine device, implantable or injectable contraceptives [i.e., Norplant or Depo-Provera] or surgical sterilization) for the duration of the study and should continue such precautions for 12 months after receiving treatment.
11. Screening physical exam must be obtained less than 7 days prior to treatment and the results must meet the following criteria:

    1. Temperature range: < 38.0 and greater and >36.0
    2. Respiratory rate: 10-20 breaths per minute
    3. Heart rate: 50 - 85 beats per minute
    4. Blood pressure: Systolic blood pressure greater than 90 mm Hg and less than 155 mm Hg
    5. % oxygen saturation by pulse oximetry: >93%
12. Screening laboratory tests will be obtained less than 7 days prior to treatment and the results must meet the following criteria:

    1. WBC > 3500/ mm3 and /or ANC > 1500/ mm3, and Platelet count 100,000/ mm3.
    2. Serum creatinine < 1.5X upper limit of normal (ULN).
    3. AST or ALT < 2.5X ULN, Alkaline phosphatase < 2.5X ULN, and Bilirubin < 1.5X ULN.
    4. INR < 1.3
    5. Hemoglobin > 10.0 g/dL
13. Negative serum pregnancy test for females of childbearing potential.
14. The patient must be capable of giving informed consent and the consent must be obtained prior to any other screening procedures that are not considered standard procedures in this patient population.
15. A baseline transthoracic echocardiogram demonstrating a left ventricular ejection fraction (LVEF) greater than 50% and no significant valvular disease (Subjects with trace or mild valvular stenosis or regurgitation will be permitted to enroll in the study).
16. Patient is able to stay within 45 minutes driving time of Johns Hopkins Hospital for 28 days following spore injection and the 7 day in-patient hospitalization period.
17. Patient is able to stay within 45 minutes driving time of Johns Hopkins Hospital for at least 35 days after recovery from all adverse events.

Exclusion Criteria -

1. Weight > 135 kg
2. Chronic renal failure requiring hemodialysis or peritoneal dialysis
3. Patients with renal cysts.
4. Tumor lesion that is not accessible to percutaneous drainage.
5. Any single contiguous lesion greater than > 12.5 cm (largest diameter).
6. The sum of the largest cross-sectional diameters from any number of non-contiguous lesions > 2 cm cannot be > 25 cm.
7. Use of any investigational drug within 30 days prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
8. Any documented evidence of primary brain malignancy or brain metastases
9. Patients with any clinically significant ascites or portosystemic hypertension, chronic jaundice or cirrhosis.
10. Patients with indwelling intrahepatic arterial pumps
11. Patients with prosthetic joints, prosthetic valves, pacemakers or any other implanted foreign materials. (non-CNS surgical clips or staples are excluded)
12. Patients with any clinically significant pleural effusions
13. Patients with any evidence of hemodynamic compromise from a pericardial effusion, circumferential pericardial effusion, or any effusion greater than 1.0 cm at any location around the heart.
14. Documented cirrhosis of the liver by clinical scenarios encompassing radiographic,clinical and laboratory results
15. Ongoing treatment with any immunosuppressive agent(s)
16. Any evidence of serious infections (such as pneumonia or pyelonephritis) or history of chronic or recurrent infectious disease in the previous 3 months.

    Less serious infections (such as acute upper respiratory tract infection(colds)or simple urinary tract infection) can be included upon the discretion of the investigator.
17. Patients with opportunistic infections, including but not limited to evidence of active cytomegalovirus, Tuberculosis, active Pneumocystis carinii, Aspergillosis,histoplasmosis, or atypical mycobacterium infection, within the previous 6 months.
18. Documented HIV infection.
19. Active or chronic Hepatitis B or Hepatitis C.
20. Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
21. History of an autoimmune disorder (eg, systemic lupus, pemphigus vulgaris,myasthenia gravis) ), requiring medication.
22. History of Diabetes Mellitus (type I or II)
23. History of rheumatic fever, endocarditis, or greater than mild valvular disease.
24. Patients who depend upon COX II inhibitors or NSAIDS
25. History of ongoing and active arterial vasculopathy (i.e. coronary artery disease, vasculitis, diabetic vasculopathy [i.e. retinopathy, nephropathy, etc.]) or evidence of end organ damage (visual loss, azotemia, and cutaneous ulcerations).
26. History of an ischemic insult in the previous 12 months (myocardial infarction, cerebra vascular accident, ischemic tissue from injury or peripheral vascular disease)
27. History of venous or lymphatic stasis resulting in venous stasis ulcers or greater than 2+ edema or lymphedema.
28. History of a significant medical illness deemed by the principal investigator or sub-investigators as unsuitable for the trial - for example:

    1. Symptomatic congestive heart failure
    2. Psychiatric Illness/Social Situation that may make study dangerous
    3. Unstable angina pectoris
29. History of a splenectomy
30. Patients with a documented Penicillin or Metronidazole allergy
31. Patients with a documented allergy to radiology contrast dye.
32. Patient with active diverticulitis
33. Patient with active dental abscesses
34. Patients with inflammatory bowel disease (IBD)
35. Women who are pregnant, lactating or breast feeding
36. Patients with angiosarcoma
37. Patients with history of a positive PPD, past TB infection or past atypical mycobacterium infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety profile, dose limiting toxicities (DLT), and maximum tolerated dose (MTD) of C. novyi-NT in humans with treatment-refractory solid tumor malignancies when given as a single intravenous injection | 2 years

SECONDARY OUTCOMES:
To document preliminary evidence of anti-tumor activity of C. novyi-NT in humans with treatment-refractory solid tumor malignancies when given as a single intravenous injection | 2 years
To analyze the pharmacokinetics of C. novyi-NT after administration to humans with treatment-refractory solid tumor malignancies when given as a single intravenous injection | 2 years
To measure the host immune and inflammatory response to C. novyi-NT in humans with treatment-refractory solid tumor malignancies when given as a single intravenous injection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Diaz, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutes, Baltimore, Maryland, United States

REFERENCES:
- [Background] Diaz LA Jr, Cheong I, Foss CA, Zhang X, Peters BA, Agrawal N, Bettegowda C, Karim B, Liu G, Khan K, Huang X, Kohli M, Dang LH, Hwang P, Vogelstein A, Garrett-Mayer E, Kobrin B, Pomper M, Zhou S, Kinzler KW, Vogelstein B, Huso DL. Pharmacologic and toxicologic evaluation of C. novyi-NT spores. Toxicol Sci. 2005 Dec;88(2):562-75. doi: 10.1093/toxsci/kfi316. Epub 2005 Sep 14. PMID 16162850
- [Background] Folkman J. A novel anti-vascular therapy for cancer. Cancer Biol Ther. 2004 Mar;3(3):338-9. doi: 10.4161/cbt.3.3.708. Epub 2004 Mar 29. No abstract available. PMID 14726666
- [Background] Dang LH, Bettegowda C, Agrawal N, Cheong I, Huso D, Frost P, Loganzo F, Greenberger L, Barkoczy J, Pettit GR, Smith AB 3rd, Gurulingappa H, Khan S, Parmigiani G, Kinzler KW, Zhou S, Vogelstein B. Targeting vascular and avascular compartments of tumors with C. novyi-NT and anti-microtubule agents. Cancer Biol Ther. 2004 Mar;3(3):326-37. doi: 10.4161/cbt.3.3.704. Epub 2004 Mar 12. PMID 14739784
- [Background] Bettegowda C, Dang LH, Abrams R, Huso DL, Dillehay L, Cheong I, Agrawal N, Borzillary S, McCaffery JM, Watson EL, Lin KS, Bunz F, Baidoo K, Pomper MG, Kinzler KW, Vogelstein B, Zhou S. Overcoming the hypoxic barrier to radiation therapy with anaerobic bacteria. Proc Natl Acad Sci U S A. 2003 Dec 9;100(25):15083-8. doi: 10.1073/pnas.2036598100. Epub 2003 Dec 1. PMID 14657371
- [Background] Dang LH, Bettegowda C, Huso DL, Kinzler KW, Vogelstein B. Combination bacteriolytic therapy for the treatment of experimental tumors. Proc Natl Acad Sci U S A. 2001 Dec 18;98(26):15155-60. doi: 10.1073/pnas.251543698. Epub 2001 Nov 27. PMID 11724950
- [Background] Agrawal N, Bettegowda C, Cheong I, Geschwind JF, Drake CG, Hipkiss EL, Tatsumi M, Dang LH, Diaz LA Jr, Pomper M, Abusedera M, Wahl RL, Kinzler KW, Zhou S, Huso DL, Vogelstein B. Bacteriolytic therapy can generate a potent immune response against experimental tumors. Proc Natl Acad Sci U S A. 2004 Oct 19;101(42):15172-7. doi: 10.1073/pnas.0406242101. Epub 2004 Oct 7. PMID 15471990
- [Background] Jain RK, Forbes NS. Can engineered bacteria help control cancer? Proc Natl Acad Sci U S A. 2001 Dec 18;98(26):14748-50. doi: 10.1073/pnas.261606598. No abstract available. PMID 11752416